CLINICAL TRIAL: NCT05098834
Title: Assessment of Lung Volumes During Liberation From Mechanical Ventilation Using Electrical Impedance Tomography in Children
Brief Title: Electrical Impedence Tomography With ENLIGHT2100
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device received FDA approval
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00108931
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Extubation
Keywords: Acute respiratory failure; Breathing tube; Mechanical ventilator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PICU and PCICU Patients (Experimental): Patients younger than 17 years of age receiving mechanical ventilation for an acute respiratory illness will be approached to participate prior to initiation of an ERT for clinical purposes.
  Interventions: Device: ENLIGHT 2100 ventilatory electrical impedance tomograph

INTERVENTIONS:
Device: ENLIGHT 2100 ventilatory electrical impedance tomograph — The ENLIGHT 2100 system will remain connected to the patient for data acquisition from immediately prior to initiation of the ERT until up to 24 hours following extubation.

SUMMARY:
Children with acute respiratory failure often need a breathing tube attached to a breathing machine, called a mechanical ventilator, to assist their breathing until they can recover. Once the cause of respiratory failure has resolved or improved enough, the breathing tube can be removed, and that is called extubation. The Extubation Readiness Test (ERT) is a simple evaluation commonly performed in the intensive care unit to determine if a child is ready to have the breathing tube removed.

The purpose of this study is to better understand how the ERT and the eventual removal of the breathing tube affect where the air is in the lungs, and whether this can help predict which children will succeed or fail having the breathing tube taken out. This can done be at the bedside with a device called electrical impedance tomograph. This novel device is painless and uses a belt fitted with sensors placed around the chest to show where the air is in the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 17 years of age admitted to the Duke Children's PICU or PCICU with acute respiratory failure due to a pulmonary illness will be considered eligible for the study

Exclusion Criteria:

* Patients with corrected gestational age less than 37 weeks
* Patients with contraindications to the ENLIGHT device (i.e. temporary or permanent pacemaker, vagal nerve stimulator, automatic implanted defibrillator, chest tubes that interfere with electrode belt placement, open chest wounds, unstable thorax, severe chest wall deformities)
* known pregnancy
* Patients previously enrolled in this study will be excluded from participation.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in expiratory lung volume as measured by global lung electrical impedance | Baseline, 60 mins, 75 mins, 90 mins

SECONDARY OUTCOMES:
Change in regional ventilation (Anterior/Posterior) distribution as measured by regional electrical impedance | Baseline, 60 mins, 75 mins, 90 mins
Change in regional ventilation (Right/Left) distribution as measured by regional electrical impedance | Baseline, 60 mins, 75 mins, 90 mins
Percent of failed extubation as measured by need for re-intubation | Within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Rotta, MD, FCCM, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No